CLINICAL TRIAL: NCT05887219
Title: Comparative Efficacy of Azelaic Acid 20% Cream Versus Hydroquinone 4% Cream as an Adjuvant to Oral Tranexamic Acid in Melasma
Brief Title: Comparison of Azelaic Acid 20 % Cream Versus Hydroquinone 4% Cream as an Adjuvant to Oral Tranexamic Acid in Melasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Zahra Nigar, Principal Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAbbottabad1987
Record Dates: First submitted 2023-05-18; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A 4 % Hydroquinone Cream Topically and Oral Tranexamic Acid (Active Comparator): Group A was managed with 4% hydroquinone cream as an adjuvant to oral tranexamic acid (250 mg twice daily)
  Interventions: Drug: Group A 4 % Hydroquinone Cream Topically and Oral Tranexamic Acid
- Group B Azelaic Acid 20 % cream for 6 months (Active Comparator): group B was managed with topical 20% azelaic acid (daily at night) for six months.
  Interventions: Drug: Group B Azelaic Acid 20 % Cream for 6 months

INTERVENTIONS:
Drug: Group A 4 % Hydroquinone Cream Topically and Oral Tranexamic Acid — Group A was managed with 4% hydroquinone cream as an adjuvant to oral tranexamic acid (250 mg twice daily) for 6 months
  Arms: Group A 4 % Hydroquinone Cream Topically and Oral Tranexamic Acid
Drug: Group B Azelaic Acid 20 % Cream for 6 months — Group B was managed with topical 20% azelaic acid (daily at night) for six months.
  Arms: Group B Azelaic Acid 20 % cream for 6 months

SUMMARY:
Methodology: Fifty female patients presented with melasma (symmetrically distributed hyperpigmented macules and patches on the face) diagnosed by consultant dermatologist on clinical presentation were included in this study. The sample size was calculated by WHO Sample Size calculator taking 31% proportion of excellent response with 4% hydroquinone as an adjuvant to oral tranexamic acid as compared to 2.25% proportion of excellent response with 20% azelaic acid, 80% power of test and 5% significance level. After randomization, patients were divided into two groups. Group A was managed with 4% hydroquinone cream as an adjuvant to oral tranexamic acid (250 mg twice daily) while group B was managed with topical 20% azelaic acid (daily at night) for six months. Clinical evaluation was done initially at the start of therapy and then at 2nd, 4th and 6th month using MASI score and patient's response. Efficacy was assessed in both groups at the end of therapy after six months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 20 to 45 years
* Presented with melasma (symmetrically distributed hyperpigmented macules and patches on the face)
* Diagnosed by consultant dermatologist on clinical presentation under wood's light.

Exclusion Criteria:

* Pregnant patients
* Women taking contraceptive pills at the time of study or past 12 months
* Any chronic illness
* Allergy to any of the agents used in the treatment
* Those taking any topical and systemic treatment for melasma in the last one month

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Melasma Area and Severity Index | 6 months
  Melasma Area and Severity Index Score was used to assess response to treatment.Lowest score=0,Highest Score 48. High score indicates worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zahra Nigar, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No